CLINICAL TRIAL: NCT05640414
Title: Healthy Families Clinic and Teaching Kitchen Program
Brief Title: Weekly Family Food Packages: Food is Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Academy of Pediatrics (Other); Ardmore Foundation (Unknown); Vitamix Foundation (Unknown)
Responsible Party: Principal Investigator, Lauren G. Fiechtner, M.D., Associate Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P002892
Record Dates: First submitted 2022-11-23; First posted 2022-12-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Food Insecurity; Overweight; Obesity; Cardiometabolic Syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Family Food Packages (Experimental)
  Interventions: Other: Weekly Family Food Packages
- Family Health Group Sessions (Experimental)
  Interventions: Other: Weekly Family Food Packages; Behavioral: Family Health Group Sessions

INTERVENTIONS:
Other: Weekly Family Food Packages — Families receive weekly family food packages for 6 months
Behavioral: Family Health Group Sessions — Families with children aged 6-17 years attend 6 monthly group sessions with cooking demonstrations
  Arms: Family Health Group Sessions

SUMMARY:
The specific aims and objectives of this proposal are to:

1. Evaluate a food pantry's weekly food distribution impact on behavioral, social and health outcomes in families.
2. In a subset of families with a child aged 6-17 years, test a pilot intervention offering the following components, with a goal of improving family behavioral, social and health outcomes:

   1. Weekly family food packages from the Revere Food Pantry
   2. 6-Monthly group sessions that include information on healthy behaviors, chronic disease management and teaching families how to prepare simple recipes based on the food they receive that week from the food pantry.

ELIGIBILITY:
Inclusion Criteria:

* Referral to the food pantry

Additional inclusion criteria for Group Sessions:

- Family has a child aged 6-17 years

Exclusion Criteria:

- Not able to speak English or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Change in BMI at 6 months | 0-6 months
  Weight in kg and height in meters will be combined to report BMI in kg/m^2, as reported in the electronic health record
Change in Food Insecurity Status at 3 months | 0-3 months
  Food insecurity status assessed by the Hunger Vital Signs questionnaire
Change in Diet Quality at 3 months | 0-3 months
  Diet quality assessed by an abbreviated food frequency questionnaire

SECONDARY OUTCOMES:
Change in Binge Eating Symptoms at 3 months | 0-3 months
  Binge eating symptoms assessed by questionnaire
Change in Blood Pressure at 6 months | 0-6 months
  Blood pressure as reported in the electronic health record
Change in Sleep at 3 months | 0-3 months
  Sleep duration as reported by questionnaire
Change in Physical Activity at 3 months | 0-3 months
  Physical activity as reported by questionnaire
Change in Screen Time at 3 months | 0-3 months
  Screen time as reported by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- MGH Revere HealthCare Center, Revere, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual-level data may be shared upon request, under the conditions that an analysis plan is prepared and approved by the PI/Co-Is, IRB approval has been obtained, and all necessary data sharing agreements have been executed.
Supporting Information: Study Protocol, ICF
Time Frame: Data can be requested by emailing the PI or Project Manager.
Access Criteria: 1. An analysis plan is prepared and approved by the PI/Co-Is,
  2. IRB approval has been obtained, and
  3. All necessary data sharing agreements have been executed.